CLINICAL TRIAL: NCT02882607
Title: Peer Groups for Healthy Pregnancy & HIV Prevention for Young Malawian Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Kamuzu College of Nursing, University of Malawi (Unknown)
Responsible Party: Principal Investigator, Kathy Norr, Professor Emerita, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01HD060461 (NIH)
Record Dates: First submitted 2016-08-01; First posted 2016-08-30 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: HIV; Pregnancy; Sexually Transmitted Infections
Keywords: HIV; Prevention; unintended pregnancy; Malawi; adolescent women; community; rural
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Reproductive Health Peer Groups
  Interventions: Behavioral: Mzanga Samala Moyo Wako ([Mzanga] Peer Groups
- Control group (No Intervention): no intervention

INTERVENTIONS:
Behavioral: Mzanga Samala Moyo Wako ([Mzanga] Peer Groups — 8 small group sessions led by community young women, focused on reproductive health, including HIV, STI and unintended pregnancy prevention; includes skill-building for self-efficacy
  Arms: Intervention group

SUMMARY:
The purpose of this study is to test the efficacy of an innovative, culturally relevant, community-based peer group intervention to increase young rural Malawian women's preconception behaviors to optimize their reproductive health. The study uses a longitudinal, two group (two-arm) design with a delayed control group.

DETAILED DESCRIPTION:
Maintaining optimal reproductive health in the context of high HIV prevalence is a serious dilemma facing young women in Malawi and other high HIV prevalence countries. Optimal reproductive health requires practicing preconception behaviors to promote overall health including avoiding HIV infection. These healthy preconception behaviors include: practicing safer sex (abstaining or using condoms) to prevent sexually transmitted infections (STIs), including HIV infection; obtaining treatment for STIs; maintaining good health habits such as diet, exercise and avoiding substance use; using an effective family planning method to prevent unintended pregnancy; and having an HIV test periodically and with the partner when conception is intended. However the Malawi Demographic and Health Survey provides evidence that few women ages 15-20 in Malawi currently practice these healthy preconception behaviors. Currently, no programs in Malawi offer an integrated approach to optimal reproductive health.

To fill this gap, this study developed an innovative, culturally relevant, community-based peer group intervention to increase young rural Malawian women's preconception behaviors to optimize their reproductive health. The intervention is called Mzanga Samala Moyo Wako ([Mzanga] Sharing Responsibility for Pregnancy Planning and HIV Prevention). Mzanga builds on the investigators' previous research in Malawi, which tested a culturally relevant HIV prevention peer group intervention that changed HIV prevention-related knowledge, attitudes, and safer sex behaviors for rural adults and adolescents. This study integrated that prior HIV prevention content with new content on maintaining health, family planning, and preconception HIV testing.

The purpose of this study is to test Mzanga's efficacy using a longitudinal, two group (two arm) design: intervention group and delayed control group. Because Mzanga is expected to diffuse widely, we randomize at the community rather than the individual level. Eighteen geographically separate rural communities stratified by size and distance from the main paved road and then randomly assigned to Mzanga or the delayed control condition. We implement Mzanga in 9 waves. A final sample of 345 per group after attrition provides adequate power (80%) to detect small-to-medium effects. After baseline data collection, the Mzanga group receives the eight-session intervention. Outcomes are measured at 9 months post-baseline (6 months post-intervention), followed by a booster session for the Mzanga group, and final evaluation at 15 months post-baseline. After the 15-month data collection, Mzanga is offered to the delayed control group.

The study aims and hypotheses are:

Aim 1. To test the efficacy of the Mzanga intervention for improving reproductive health outcome mediating and behavioral variables for Malawian rural young women at 9 and 15 months post-baseline.

H1.Controlling for baseline differences and group effects, compared to the delayed control group, the intervention group will show more positive mediating and behavioral outcomes:

1. Practice safer sex,
2. Obtain prompt treatment for STI symptoms;
3. Maintain good health habits (diet, exercise, substance use);
4. Use an effective family planning method except when pregnancy is intended;
5. Have an HIV test periodically, with partner when conception is intended; and
6. More positive scores for the mediating variables of knowledge, attitudes, perceived norms, self-efficacy, and intentions for each of these behaviors.

Aim 2. To test a theoretical model of the mechanisms through which the Mzanga intervention changes preconception health behaviors of young women in rural Malawi.

H2. Mzanga's effects on healthy preconception behaviors (a-e above) will be mediated by knowledge, attitudes, perceived norms, self-efficacy, and intention scores.

ELIGIBILITY:
Inclusion Criteria:

* lives in designated community

Exclusion Criteria:

* cognitive or other condition that makes the participant unable to converse in a group or answer questions

Ages: 15 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 810 (Actual)
Dates: Start 2009-05; Primary Completion 2014-07 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
change in unprotected sex | Change from baseline to 15 months post-baseline
  Change in having sex without a condom (n the last 2 months) from baseline to 15-months post-baseline, measured by 2 questions, have you had sex in the last 2 months, and (for those who had sex) have you used a condom 'always, sometimes or never'; if had sex and have not used a condom always are coded 'yes', had unprotected sex; all other responses are coded no.

SECONDARY OUTCOMES:
Change in having had an HIV test | Change in having had an HIV test from baseline to 15 months post-baseline
  change in whether had a recent HIV test (within the last 12 months) from baseline to 15-months post-baseline
change in having sexually transmitted infection (STI) symptoms | baseline to 15 months post-baseline
  change in reported STI symptoms between baseline and 9-month and 15-month survey
Change in unintended pregnancy | Change in unintended pregnancy from baseline to 15 months post-intervention
  Change in reported unintended pregnancy between baseline and 15-months post-baseline; measured by whether pregnant, confirmed visually and by pregnancy test, and whether reported in intending to become pregnant

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen F. Norr, PhD, Principal Investigator — University of Illinois at Chicago

IPD SHARING:
Plan to Share IPD: No
Deidentified data will be made available 5 yrs. after study completion by request to the PI